CLINICAL TRIAL: NCT06399822
Title: Impact of Capillaroscopy on the Management of Undifferentiated Connective Tissue Disease: a Randomized Pilot Clinical Study
Brief Title: Impact of Capillaroscopy on the Management of Undifferentiated Connective Tissue Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-7303
Record Dates: First submitted 2024-04-22; First posted 2024-05-06 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Undifferentiated Connective Tissue Diseases
Keywords: undifferentiated connective tissue disease; capillaroscopy; randomized pilot clinical study
MeSH Terms: conditions — Undifferentiated Connective Tissue Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capillaroscopy (Active Comparator): In the capillaroscopy group, the capillaroscopy will be performed in the month following recruitment.
  Interventions: Diagnostic Test: Nail capillaroscopy
- Control (Other): In the control group, the capillaroscopy will be performed six months (+/- 2 weeks) after recruitment.
  Interventions: Diagnostic Test: Nail capillaroscopy

INTERVENTIONS:
Diagnostic Test: Nail capillaroscopy — The intervention studied as part of the project is capillaroscopy. This examination consists of visualizing the capillaries located at the base of the nail using a device called a capillaroscope. This device magnifies the image of the capillaries to clearly visualize them. Capillaries are the smallest blood vessels, which allow the passage of only one red blood cell at a time. At the nail bed, they form a network of loops and are aligned next to each other. This alignment allows them to be viewed over their entire length. Researchers have described abnormalities in capillaries that are associated with certain diseases involving microvascular damage.
  The results of capillaroscopy will be reported qualitatively, for all eight long fingers examined.

SUMMARY:
Connective tissue diseases (CTD) are a group of diseases with diverse manifestations, most often multisystemic, which share an autoimmune etiology. They include Systemic lupus erythematosus (SLE), Systemic sclerosis (SSc), Sjögren's syndrome (SS), Inflammatory myopathies (IM) and Mixed connective tissue disease (MCTD).

Many patients in rheumatology present signs and symptoms of CTD, but without meeting all the classification criteria for one of these diseases. These patients will generally receive a diagnosis of undifferentiated connective tissue disease (UCTD). It is increasingly suggested that there are two subgroups of patients with UCTD: one which will eventually evolve into a better characterized CTD (approximately 30% of patients at 5 years) and another with a more benign prognosis. The optimal management of patients with UCTD is not clearly established.

Capillaroscopy is a diagnostic test used in the investigation of patients with CTD. It is a low-cost, non-invasive, rapid and specific test in the evaluation of this class of diseases. Its role is now well established in the diagnosis of SSc and in the investigation of Raynaud's phenomenon. In addition, capillaroscopy helps to identify patients suffering from CTD more quickly.

Knowledge about the role of capillaroscopy in UCTD is more limited. It is established that a significant proportion of patients with UCTD present abnormalities on UCTD present non-specific abnormalities and 11% present a scleroderma pattern. In these patients, abnormal capillaroscopy seems to increase the risk of progressing to a better characterized CTD, notably SSc.

However, although capillaroscopy is increasingly used in rheumatology in patients with CTD, more research is needed to clarify the role of this examination in UCTD. First, it is not established whether capillaroscopy should be performed in all patients with UCTD, nor when exactly it should be performed. There also remain questions about the impact of capillaroscopy on the prognosis and management of patients with this disease. To our knowledge, there is no prospective study that has addressed this question. The investigators hypothesize that in patients with UCTD, capillaroscopy compared to usual care makes it possible to increase the proportion of patients obtaining a diagnosis of better characterized CTD in the first six months of follow-up.

DETAILED DESCRIPTION:
This is a pilot randomized controlled clinical trial. This monocentric project will be carried out within the rheumatology department of the Quebec university hospital.

The main objective of the project is to determine, in patients with undifferentiated connective tissue disease, to what extent capillaroscopy compared to usual care influences the proportion of patients obtaining a diagnosis of better characterized connective tissue disease in the first six months of follow-up.

The secondary objectives are:

1. Determine, in patients with undifferentiated connective tissue disease, to what extent capillaroscopy influences the following factors after capillaroscopy:

   * The proportion of patients obtaining a diagnosis of better characterized connective tissue disease at 12 months;
   * Medication changes (addition, discontinuation or change in dosage of non-biological disease modifying drugs, biological disease modifying drugs, medications for Raynaud's syndrome and corticosteroids) at 6 and 12 months;
   * The number of medical visits in rheumatology, medical visits in specialties other than rheumatology, hospitalizations and emergency medical visits at 6 and 12 months;
   * The number of additional examinations (blood samples, radiological examinations or others) carried out which were prescribed by the treating rheumatologist at 6 and 12 months;
   * A change in lifestyle habits (smoking, alcohol and drug consumption, physical activity, diet) at 6 and 12 months;
   * Patients' quality of life assessed by the health assessment questionnaire, short form survey-36 and Patient-Reported Outcomes Measurement Information System-29 questionnaires at 6 and 12 months;
   * Patient acceptability and satisfaction with the intervention under study at 12 months;
2. Evaluate the feasibility of recruiting participants in this study (the investigators will measure the number, proportions and rates of patients recruited and retained, as well as the number of individuals screened, eligible and recruited).

The investigators will recruit 40 patients with a diagnosis of undifferentiated connective tissue disease and referred for a capillaroscopy examination in rheumatology as part of clinical practice.

Once recruited, participants will be randomized into two groups, in a 1:1 ratio, stratifying for gender and duration since the onset of the first symptoms of the disease (less than three years and three years and more). The randomization blocks will be generated by the biostatistician.

In the intervention group, a capillaroscopy will be performed in the month following recruitment. In the control group, capillaroscopy will be performed six months (+/- two weeks) after recruitment.

The intervention studied as part of the project is capillaroscopy. This examination consists of visualizing the capillaries located at the base of the nail using a device called a capillaroscope. This device magnifies the image of the capillaries to clearly visualize them. Capillaries are the smallest blood vessels, which allow the passage of only one red blood cell at a time. At the nail bed, they form a network of loops and are aligned next to each other. This alignment allows them to be viewed over their entire length. Researchers have described abnormalities in capillaries that are associated with certain diseases involving microvascular damage.

Participants will be invited to attend an appointment at the outpatient clinic to perform the capillaroscopy. The date of this appointment will depend on the group into which they have been randomized. If they are assigned to the intervention group, capillaroscopy will be performed within one month after inclusion in the study. If they are assigned to the control group, capillaroscopy will be performed six months after inclusion in the study, (+/- two weeks). If the capillaroscopy appointment is missed, a new appointment will be scheduled within two weeks.

The results of capillaroscopy will be reported qualitatively, for all eight long fingers examined. This approach was chosen since it best represents current clinical practice. The capillaroscopy results will therefore be classified into one of the following categories: normal; nonspecific changes; scleroderma pattern; non-diagnostic quality.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 and over;
* Have been diagnosed with undifferentiated connective tissue disease by a rheumatologist;
* Meet the preliminary classification criteria for undifferentiated connective tissue disease: present signs and symptoms suggestive of connective tissue disease, but do not meet the criteria for a connective tissue disease and have a positive antinuclear antibody on at least 2 occasions;
* Have developed the first signs and symptoms of the disease less than 10 years before recruitment.

Exclusion Criteria:

* In the opinion of the clinician, have a health condition that does not allow a delay of six months before carrying out the capillaroscopy;
* Have been diagnosed and/or meet the classification criteria for another connective tissue disease (for example, systemic lupus, etc.);
* Have already performed a capillaroscopy in the past, regardless of the time or the reason;
* Be unable to consent or respond to questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who transitioned from a diagnosis of undifferentiated connective tissue disease to a diagnosis of better characterized connective tissue disease | 6 months
  The primary endpoint of the study will be the proportion of participants who transitioned from a diagnosis of undifferentiated connective tissue disease to a diagnosis of better characterized connective tissue disease at 6 months.

SECONDARY OUTCOMES:
Proportion of participants who went from a diagnosis of undifferentiated connective tissue disease to a diagnosis of better characterized connective tissue disease | 12 months
  The proportion of participants who went from a diagnosis of undifferentiated connective tissue disease to a diagnosis of better characterized connective tissue disease at 12 months;
Proportion of participants with a medication change from the baseline visit | 6 and 12 months
  The proportion of participants with a medication change from the baseline visit (defined as the addition, discontinuation, or dosage change of nonbiologic disease-modifying drugs, biologic disease-modifying drugs, Raynaud's medications, and corticosteroids) at 6 and 12 months
Average number of rheumatology medical visits per participant | 6 and 12 months
  The average number of rheumatology medical visits per participant at 6 and 12 months (continuous value);
Average number of medical visits in specialties other than rheumatology per participant | 6 and 12 months
  The average number of medical visits in specialties other than rheumatology per participant at 6 and 12 months (continuous value);
Average number of hospitalizations per participant | 6 and 12 months
  The average number of hospitalizations per participant at 6 and 12 months (continuous value);
Average number of emergency room visits per participant | 6 and 12 months
  The average number of emergency room visits per participant at 6 and 12 months (continuous value);
Average number of additional examinations | 6 and 12 months
  The average number of additional examinations (blood samples, radiological examinations or others) which were prescribed by the treating rheumatologist per participant at 6 and 12 months (continuous value);
Proportion of patients with a healthy weight | 6 and 12 months
  The proportion of patients with a healthy weight (body mass index of 18.5 to 24.9);
Average number of alcohol drinks (standard drinks) consumed per week and per participant | 6 and 12 months
  The average number of alcohol drinks (standard drinks) consumed per week and per participant at 6 and 12 months (continuous value);
Proportion of patients who are active smokers, former smokers and have never smoked | 6 and 12 months
  Smoking status (i.e. the proportion of patients who are active smokers, former smokers and have never smoked) at 6 and 12 months;
Average number of cigarettes smoked per day per participant | 6 and 12 months
  The average number of cigarettes smoked per day per participant at 6 and 12 months (continuous value);
Proportion of participants using tobacco products other than cigarettes | 6 and 12 months
  The proportion of participants using tobacco products other than cigarettes at 6 and 12 months;
Proportion of participants using cannabis products | 6 and 12 months
  The proportion of participants using cannabis products at 6 and 12 months;
Proportion of participants using drugs other than cannabis | 6 and 12 months
  The proportion of participants using drugs other than cannabis at 6 and 12 months;
Average number of minutes of moderate to high intensity aerobic physical activity performed per week and per participant | 6 and 12 months
  The average number of minutes of moderate to high intensity aerobic physical activity performed per week and per participant at 6 and 12 months (continuous value);
Proportion of participants who reported adopting a diet following the healthy eating recommendations of Canada's Food Guide | 6 and 12 months
  The proportion of participants who reported adopting a diet following the healthy eating recommendations of Canada's Food Guide at 6 and 12 months.
Average score on the Health Assessment Questionnaire | 6 and 12 months
  The average score on the Health Assessment Questionnaire (from 0 to 3, with 3 decimal places);
Average score for the eight components of the Short form survey 36 questionnaire | 6 and 12 months
  The average score for the eight components of the short form survey 36 questionnaire (from 0 to 100, with 2 decimal places): (1) physical functioning, (2) role limitations due to physical health problems, (3) bodily pain, (4) general health perceptions, (5) energy/fatigue, (6) social functioning, (7) role limitations due to personal or emotional problems and (8) emotional well-being;
Average score on the eight components of the Patient-Reported Outcomes Measurement Information System29 scale | 6 and 12 months
  The average score on the eight components of the Patient-Reported Outcomes Measurement Information System29 scale (without decimal): (1) physical function (4 to 20), (2) anxiety (4 to 20), (3) depression (4 to 20), (4) fatigue (4 to 20), (5) sleep disturbances (4 to 20), (6) ability to participate in social roles and activities (4 to 20), (7) ) pain interference (4 to 20) and (8) pain intensity (0 to 10).

OTHER OUTCOMES:
Questionnaire of acceptability of capillaroscopy | 6 and 12 months
  The investigators will determine the acceptability of capillaroscopy by a questionnaire consisting in 4 questions (duration of capillaroscopy, absence of pain and discomfort, acceptability of capillaroscopy to investigate the participant condition, recommendation of capillaroscopy to somebody else) to be answered by the use of 5-point Likert scale (from totally agree to totally disagree).
Questionnaire of satisfaction about study questionnaires | 6 and 12 months
  The investigators will evaluate the satisfaction of participants about study questionnaires by a questionnaire consisting in two questions (easiness to understand questionnaires, adequateness of time to complete questionnaires) to be answered by the use of 5-point Likert scale (from totally agree to totally disagree).
Number of individuals screened, eligible and recruited. | 6 and 12 months
  The investigators will measure the number of individuals screened, eligible and finally recruited in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia Michou, MD PhD, Principal Investigator — CHU de Quebec (Université Laval)
Locations (1):
- CHU de Quebec-Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The established and evolving role of nailfold capillaroscopy in connective-tissue disease — https://www.intechopen.com/chapters/65046